CLINICAL TRIAL: NCT04770259
Title: Generation of a Pre-surgical Conditioning Protocol for Frail Elderly People in Order to Reduce Hospitalization Days.
Brief Title: Pre-surgical Protocol for Frail Elderly People in Order to Reduce Hospitalization Days (APOPM).
Acronym: APOPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Victor Contreras, MSN, Research associate, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200302001
Record Dates: First submitted 2021-02-15; First posted 2021-02-25 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Surgery; Old Age; Debility; Frail Elderly Syndrome; Post-Operative Confusion; Older Adults; Perioperative Care; Urologic Diseases; Digestive Disease; Anesthesia; Nurse-Patient Relations
Keywords: Older adults; Perioperative Care; Frail Elderly Syndrome; Pre-habilitation; length of stay in hospital
MeSH Terms: conditions — Frailty; Urologic Diseases; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: randomized controlled, longitudinal.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will have a nursing evaluation and then follow the surgeon's instructions in the current standard way until de surgery day. In that day the RN will be evaluate again these group. Then, this group will be followed within the hospital and the first, second and third month after discharge.
- Intervention (Experimental): The intervention group will have a nursing evaluation and then will attend an evaluation by geriatarics team, kinesiology and nutrition, where a plan of physical cardiovascular, nutritional and metabolic prehabilitation is delivered. On the day of surgery, the RN will evaluate this group again. Then, this group will be followed within the hospital and the first, second and third month after discharge.
  Interventions: Other: Timely pre-surgical conditioning

INTERVENTIONS:
Other: Timely pre-surgical conditioning — Timely pre-surgical conditioning seeks to prepare frail, pre-frail and / or dependent older patients for the surgery process. For which a work plan has been designed according to your needs and health conditions.
  Arms: Intervention

SUMMARY:
Elderly people (EP) have increased, as well as life expectancy at birth. In Chile there are more than 2 million 800 thousand EP, which corresponds to 1/6 of the Chilean population.

The EP have a higher disease burden and mortality when facing surgery and in the postoperative period.

Thus, this population frequently has longer hospital stays due to its degree of fragility, surgical complications or decompensation of its underlying pathologies, directly affecting health care systems.

An inadequate preparation of the EP prior to surgery determined that the requirements of in-hospital as well as out-of-hospital care are extended, with the consequent which entails a higher cost in health.

Current research underestimates the conditions of frailty and dependence in the EP. In addition, it is not routinely evaluated prior to surgery, as well as nutritional, metabolic, cognitive status and / or delirium screening is performed.

There are accelerated recovery programs, which relate their interventions to specific pathologies; however, the age of the person is not taken into account.

Surgical pre-habilitation interventions in the EP usually focus their efforts on physical and cardiovascular aspects, not including an integrative pre-surgical evaluation.

Based on the foregoing, a prospective, interventional, longitudinal and randomized study has been proposed in a population of the EP who will undergo elective urology and coloproctology surgeries in two university hospitals (private and public).

The objective of this study is to evaluate how the implementation of a timely pre-surgical conditioning (APO) protocol for frail elderly people reduces the days of hospital stay.

The APO considers the most relevant aspects of physical and cardiovascular pre-habilitation, in addition to contemplating evaluations of frailty, dependence, cognitive status, screening for delirium, nutritional and metabolic.

DETAILED DESCRIPTION:
A prospective, interventional, longitudinal and randomized study has been proposed in a population of the EP who will undergo elective urology and coloproctology surgeries in two university hospitals: Red de Salud UC-Christus and Hospital Clinico La Florida. Both based on Santiago de Chile.

The objective of this study is to evaluate how the implementation of a timely pre-surgical conditioning (APO) protocol for frail elderly people reduces the days of hospital stay.

PM will be screened according to: co-morbidities, degree of frailty and dependence. This procedure will be carried out by a trained register nurse (RN) from the team at each center, who through a random system will enter 50% of the patients to the APO protocol (intervention) and the other 50% to the standard protocol of each institution. After that the RN will measure nutritional and cognitive status, drugs and alcohol consume and will take the protocol blood samples in the first evaluation two to three days after receiving an order for surgery for the physician.

The APO considers the evaluations for a geriatric team, physical therapist team and nutritionist team in order to find out the most relevant aspects of physical, cardiovascular geriatric syndromes, cognitive status, nutritional and metabolic status.

physical therapist team and nutritionist team they will prepare to the EP to surgery with physical, cardiovascular and dietary protocols adjusted to the patient, for the time of 4 to 5 weeks before surgery.

Upon admission of hospitalization for surgery, the RN in each of the two hospitals will evaluate the state of frail and dependence, nutritional and cognitive status, drugs and alcohol consume and delirium status in which the patients of both groups arrive.

The analgesia and anesthesia of all patients in both groups, control and intervention, will be standardized to reduce confounding associated with intra- and postoperative anesthesia and analgesia.

The registered nurse will follow the patient throughout the in-hospital process and via telemedicine or face-to-face will interview patients one month, second month and third month after discharge in search of possible problems associated with the peri-operative process.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery of urology and / or minimally invasive coloproctology under general anesthesia
* Pre-frail, frail patients.
* Patients with a moderate to severe degree of dependence

Exclusion Criteria:

* Emergency surgery patients.
* Patients who are hospitalized prior to surgery for urgent reasons and / or complications from another surgery.
* Patients diagnosed with delirum, dementia or similar mental illness.

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Average of 5 to Days of hospital stay until discharge after surgery
  Reduction of length of hospital stay in terms of days after surgery of frail elderly enrolled in the control and intervention arm.
Change of the degree of the frailty in the elderly patients during the perioperative process | One month before surgery, the 1 day of the surgery up to 3 months after discharge.
  Change from Baseline in the degree of preoperative frailty in the elderly patients in both arms with Frail Scale 0= Robust, 1= Pre - Frail, 3-5 = Frail; Fried phenotype of frailty 0= Robust, 1= Pre - Frail, 3-5 = Frail and Clinical Frail Scale 1 to 9, 1 is very fit and 9 is a terminal patients.
Change of the nutritional and metabolic status in the elderly patients during the perioperative process | One month before surgery, the 1 day of the surgery up to 3 months after discharge.
  Change from Baseline in the nutritional and metabolic status in the in the elderly patients in both arms measure with the Mini Nutritional Assessment scale.
  12-14 points: Normal nutritional status 8-11 points: At risk of malnutrition 0-7 points: Malnourished
Assessment functional independence in the elderly patients preoperative and postoperative | One month before surgery, the 1 day of the surgery up to 3 months after discharge.
  Assessment functional independence with the Barthel Index for Activities of Daily Living. 0 to 100. 0 is Totally dependent and 100 totally independent
Change of the cardiorespiratory and muscular system in the elderly patients during the perioperative process | One month before surgery, the 1 day of the after surgery up to 3 days post surgery.
  Change from Baseline of the cardiorespiratory and muscular system in the elderly patients before and after surgery with Short Physical Performance Battery (Score 0 - 12, 0 = lower physical performance and 12 = higher physical performance); 6 Minute Walk Test (ranges from 400 to 700 m, the main predictor variables being gender, age and height) or 2 minute step Test (record the total number of times the right knee reaches the tape level in two minutes. The recommended ranges for this test based on age groups from Jones & Rikli, 2002).

SECONDARY OUTCOMES:
Change of the cognitive state in the elderly patients during the perioperative process | One month before surgery, the 1 day of the surgery up to 3 months after discharge.
  Change of the cognitive state in the elderly patients during the perioperative process with Mini Cog test (0-2 points indicates positive screen for dementia and 3-5 points indicates negative screen for dementia); AD8 (0 to 8, and over 2 is positive for dementia), and/or MoCA test (scores range between 0 and 30. A score of 26 or over is considered to be normal).
Identify the appearance during the perioperative process of the delirum in the elderly patients | 1 day before surgery and every day every 12 hours post surgery until discharge
  Identify the appearance during the perioperative process of the delirum in the elderly patients with Confusion assessment method (CAM), CAM=negative is delirium absent and CAM=positive is delirum present, the same for CAM-Intensive Care Unit (CAM-ICU) CAM-ICU=negative is delirium absent and CAM-ICU=positive is delirum present.
Identify morbidity and post-operative complications | Identify morbidity and mortality and post-operative complications one, two and three month after surgery discharge
  Identify post-operative complications with Claven-Dindo classification. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V).
Identify the mortality post-operative | One, two and three month after surgery discharge
  Identify the mortality post-operative in the frail elderly enrolled in the controls and intervention arm.
  Proportion of deaths from a certain of frail elderly patients after surgery compared to the total number of elderly people after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Elgueta, MD, Principal Investigator — Assistant Profesor
Locations (2):
- Chile (2):
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Hospital de La Florida, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Yes
Timely pre-surgical conditioning protocol for frail older people.
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: Certificate letter or institucional e-mail

REFERENCES:
- [Background] Edelmuth SVCL, Sorio GN, Sprovieri FAA, Gali JC, Peron SF. Comorbidities, clinical intercurrences, and factors associated with mortality in elderly patients admitted for a hip fracture. Rev Bras Ortop. 2018 Aug 2;53(5):543-551. doi: 10.1016/j.rboe.2018.07.014. eCollection 2018 Sep-Oct. PMID 30245992
- [Background] Bolliger M, Kroehnert JA, Molineus F, Kandioler D, Schindl M, Riss P. Experiences with the standardized classification of surgical complications (Clavien-Dindo) in general surgery patients. Eur Surg. 2018;50(6):256-261. doi: 10.1007/s10353-018-0551-z. Epub 2018 Jul 24. PMID 30546385
- [Background] Beggs T, Sepehri A, Szwajcer A, Tangri N, Arora RC. Frailty and perioperative outcomes: a narrative review. Can J Anaesth. 2015 Feb;62(2):143-57. doi: 10.1007/s12630-014-0273-z. Epub 2014 Nov 25. PMID 25420470
- [Background] Ferris DK, Willet-Brown J, Martensen T, Farrar WL. Interleukin 3 stimulation of tyrosine kinase activity in FDC-P1 cells. Biochem Biophys Res Commun. 1988 Aug 15;154(3):991-6. doi: 10.1016/0006-291x(88)90237-9. PMID 3261586
- [Derived] Contreras V, Elgueta MF, Balde D, Astaburuaga P, Carrasco M, Pedemonte JC, Nicoletti MN, Medina Diaz R, Franco S, Agurto R, Vivanco C, Figueroa C, Alamos M, Cuzmar Benitez V, Vargas B, Barraza B, Rematal C, Cortinez LI. Prehabilitation for Chilean frail elderly people - pre-surgical conditioning protocol - to reduce the length of stay: randomized control trial. Minerva Anestesiol. 2024 Dec;90(12):1098-1107. doi: 10.23736/S0375-9393.24.18245-4. PMID 39836361